CLINICAL TRIAL: NCT05577455
Title: Non-inferiority Randomized Controlled Study on Kidney Tonifying and Blood Circulation Regulating Therapy (Bu Shen Tiao Xue) of Different Intervention Courses in Improving IVF-ET Pregnancy Outcomes in DOR Patients
Brief Title: Efficacy of Traditional Chinese Medicine on Ameliorating IVF-ET Outcomes of Diminished Ovarian Reserve Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00006761-M2022270
Record Dates: First submitted 2022-10-09; First posted 2022-10-13 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-09

CONDITIONS: Diminished Ovarian Reserve; Infertility, Female
Keywords: traditional Chinese medicine; in vitro fertilization and embryo transfer; diminished ovarian reserve
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Intervention Model Description: After the patients complete the relevant examinations, and those who meet the inclusion criteria sign the informed consent, they are sequentially assigned to two groups according to the randomization table. The intervention begins from the second menstrual cycle prior to IVF-ET in the experimental group and third menstrual cycle prior to IVF-ET in the control group. TCM treatment is initiated on the 5th day of menstruation in both groups, and medical prescriptions before and after ovulation are administered successively. Subjects do not take any medicine on the 1st to 4th day of menstruation and medications are discontinued on the day of HCG. The TCM is decocted by our hospital, and patients are instructed to take one dose of the the decoction warm per day (400 ml per dose) one hour after meals twice (once in the morning and once in the evening). The occurrence of spontaneous pregnancy and adverse reactions are recorded and dealt with promptly throughout the drug application period.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- administration for 2 menstrual cycles group (Experimental): This group will receive TCM treatment before 2 menstrual cycles of IVF-ET.
  Interventions: Drug: Medical prescription before ovulation; Drug: Medical prescription after ovulation
- administration for 3 menstrual cycles group (Active Comparator): This group will receive TCM treatment before 3 menstrual cycles of IVF-ET.
  Interventions: Drug: Medical prescription before ovulation; Drug: Medical prescription after ovulation

INTERVENTIONS:
Drug: Medical prescription before ovulation — Medical prescription before ovulation, modified two solstices pill and Si-Wu-Tang: 15g of Nv Zhen Zi (Fructus Ligustri Lucidi), 10g of Mo Han Lian (Yerbadetajo herb), 15g of Gou Qi Zi (Fructus lycii), 20g of Tu Si Zi (Semen cuscutae), 15g of Shu Di (Radix Rehmanniae Preparata), 10g of Dang Gui (Angelica sinensis), 10g of Bai Shao (Paeonia lactiflora Pallas), 20g of Sheng Shan Yao (Rhizoma Dioscoreae), 15g of Fu Pen Zi (Raspberry), and 15g of Shan Yu Rou (Fructus corni). The medical prescription is initiated on the fifth day of menstruation and is taken continuously for 10-15 days.
Drug: Medical prescription after ovulation — Medical prescription after ovulation, modified Er Xian decoction for promoting fertilization and Si-Wu-Tang: 10g of Xian Mao (Curculigo orchioides), 15g of Xian Ling Pi (Epimedium Herb), 15g of Ba Ji Tian (Morinda officinalis), 20g of Tu Si Zi (Semen cuscutae), 15g of Nv Zhen Zi (Fructus Ligustri Lucidi), 15g of Zi Shi Ying (Fluoritum), 15g of Shu Di (Radix Rehmanniae Preparata), 10g of Dang Gui (Angelica sinensis), 10g of Bai Shao (Paeonia lactiflora Pallas), and 10g of Chuan Xiong (Szechwan Lovage Rhizome). The medical prescription is administered continuously for 10-15 days after ovulation, based on follicle development and endometrial growth monitored by ultrasound.

SUMMARY:
Patients with diminished ovarian reserve (DOR) who undergo in vitro fertilization and embryo transfer (IVF-ET) are included as the research subjects. The effects of Traditional Chinese Medicine (TCM) for kidney tonifying and blood circulation regulating of different intervention courses on ovarian hyporesponsiveness, IVF-ET outcome and clinical compliance in DOR patients are studied by a non-inferiority randomized controlled trial. The purpose is to identify the breakthrough point and treatment timing of TCM treatment, explore the best treatment course of TCM, and optimize the TCM therapeutic regimen.

DETAILED DESCRIPTION:
IVF-ET is one of the major techniques to treat infertility in DOR patients, but poor ovarian response and low pregnancy rate have been the bottleneck problems. China has original advantages in Traditional Chinese Medicine (TCM) treatment. The kidney tonifying and blood circulation regulating therapy is a pre-IVF-ET intervention treatment characterized by sequential treatment according to menstrual cycle formed in the previous investigations by the research group. It can ameliorate ovarian hyporesponsiveness and improve the success rate of IVF-ET, but the compliance is poor due to the long intervention course. Identifying the time point of TCM intervention to further optimize the treatment plan is the key to improving the pregnancy rate. Therefore, DOR patients who receive IVF-ET are enrolled as the research objects in this project, who are divided into the experimental group and control group with a randomized controlled non-inferiority design, and receive sequential TCM therapy for kidney tonifying and blood circulation regulating from the fifth day of menstruation at the second menstrual cycle and the third menstrual cycle prior to IVF-ET, respectively, until the day of human chorionic gonadotrophin (hCG) administration. The number of oocytes retrieved, the rate of high-quality embryos, the dosage and administration days of Gn, the levels of estradiol (E2) and progesterone (P) and the clinical pregnancy rate on hCG day are compared between the two groups. Meanwhile, the compliance of patients in the two groups with different treatment regimens is compared. This project aims to verify that the efficacy of the treatment plan implemented from the second menstrual cycle prior to IVF-ET may not be inferior to that from the third menstrual cycle prior to IVF-ET on improving the pregnancy outcomes of DOR patients, while the compliance is better. The results of the study will provide a reference basis for the precise treatment of TCM prior to IVF-ET.

ELIGIBILITY:
Inclusion Criteria:

1. Female, 20 years old ≤ age ≤ 42 years old;
2. The menstrual cycle is generally regular; 21 days < menstrual cycle < 35 days;
3. Those who meet the diagnostic criteria for DOR in Western medicine;
4. Those who meet the TCM differential criteria of kidney deficiency syndrome;
5. Those who are scheduled to undergo IVF-ET;
6. Those who voluntarily participate in this clinical trial and sign a written informed consent.

Exclusion Criteria:

1. Those who have a history of two or more spontaneous abortions (excluding biochemical pregnancy abortion) or three or more previous transplantations without achieving clinical pregnancy;
2. Those who have premature ovarian failure or ovarian gonadotropin resistance syndrome;
3. Those who have untreated uterine malformation or abnormality: double uterus, septate uterus (complete or incomplete);
4. Those who have untreated unilateral or bilateral hydrosalpinx;
5. Those who have uncured endometrial diseases (such as endometritis, endometrial polyps, endometriosis), adenomyosis, intrauterine adhesions, etc., and those with uterine fibroids of more than 4 cm;
6. Those who have endocrine diseases such as polycystic ovary syndrome, hyperprolactinemia, hyperandrogenism, hypothyroidism, abnormal adrenal function, etc., which affect ovulation;
7. Infertile patients with abnormal ovarian function caused by immunological factors, genetic factors or congenital physiological defects;
8. Those who have received pelvic radiotherapy;
9. Those who are known or suspected of having sex hormone-related malignant tumors;
10. Those who are allergic or intolerable to the medications involved in the study;
11. Those with contraindications to assisted reproductive technology or pregnancy, such as uncontrolled abnormal liver and renal function, diabetes, hypertension, thyroid disease, symptomatic heart disease, moderate to severe anemia, history of malignant tumor or history of thromboembolism or thrombosis formation tendency, serious mental illness, acute infection of urogenital system, sexually transmitted disease, extremely bad habits such as drug use, exposure to teratogenic radiation, poison, drugs (such as prednisone and other hormones, epinephrine, antibiotics, antihypertensive drugs, cardiovascular and cerebrovascular drugs, antiviral drugs) and are still under the effect of the drugs; and those whose uterus is unable to perform the function of pregnancy or who are intolerant of pregnancy due to physical diseases during pregnancy;
12. Those who have taken other TCMs or proprietary Chinese medicines that can invigorate the kidney or affect the evaluation of drug efficacy in the past 30 days;
13. Other patients who are deemed unsuitable to participate in this study by the researchers;
14. Those who are participating in other clinical trials;
15. Those who do not agree to participate in this study or do not sign the informed consent form.

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 266 (Estimated)
Dates: Start 2022-11-10 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of oocytes retrieved | up to 15 weeks from enrollment
  The number of oocytes retrieved by puncture under the guidance of vaginal ultrasound

SECONDARY OUTCOMES:
High-quality embryo rate (%) | up to 15 weeks from enrollment
  Number of high-quality embryos / the total number of normal cleavage embryos × 100%
Clinical pregnancy rate | up to 15 weeks from enrollment
  Ultrasound monitoring is performed 30 days after embryo transfer
Compliance with the treatment plan | up to 15 weeks from enrollment
  The situation of continuous treatment of the research subjects is recorded; the compliance of the experimental group = the number of cases who receive continuous treatment for 2 months / the total number of patients in the experimental group; the compliance of the control group = the number of cases who receive continuous treatment for 3 months / the total number of patients in the control group
Gonadotrophin (Gn) administration day | up to 15 weeks from enrollment
  Record the total gonadotrophin (Gn) administration day
Gn dosage | up to 15 weeks from enrollment
  Record the average dose of Gn administration
Levels of LH | up to 15 weeks from enrollment
  Obtained by blood sampling
Levels of E2 | up to 15 weeks from enrollment
  Obtained by blood sampling
Levels of P | up to 15 weeks from enrollment
  Obtained by blood sampling
Antral follicle count (AFC) | up to 15 weeks from enrollment
  Changes of AFC before and after TCM intervention
Levels of FSH | up to 15 weeks from enrollment
  Obtained by blood sampling
Levels of AMH | up to 15 weeks from enrollment
  Obtained by blood sampling
Health economics indicators | up to 15 weeks from enrollment
  Average daily cost and total cost

CONTACTS AND LOCATIONS:
Overall Officials: Dong Li, Study Chair — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No